CLINICAL TRIAL: NCT00054301
Title: Intraoperative Radiation Therapy to the Tumor Bed for Boost Treatment After Lumpectomy Prior to Whole Breast Radiation in Breast Conservation Candidates
Brief Title: Radiation Therapy After Lumpectomy in Treating Women With Ductal Carcinoma in Situ or Invasive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Shelli Hanks, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICC4102
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: adjuvant therapy
Procedure: conventional surgery — Patients undergo excisional biopsy or surgery.
Radiation: intraoperative radiation therapy — Patients undergo excisional biopsy or surgery followed by an intraoperative dose of radiation to the tumor cavity.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation during surgery followed by external-beam radiation to the entire breast may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of radiation therapy during surgery followed by whole-breast radiation therapy in treating women who have undergone lumpectomy for ductal carcinoma in situ or invasive breast cancer

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of intraoperative radiotherapy boost to the tumor bed on acute complications after lumpectomy (before whole breast irradiation) in women with ductal carcinoma in situ or invasive adenocarcinoma of the breast.
* Determine the local recurrence rates in patients treated with this regimen.
* Determine the cosmetic outcome in patients treated with this regimen.

OUTLINE: Patients undergo excisional biopsy or surgery followed by an intraoperative dose of radiation to the tumor cavity. Postoperatively, patients undergo external beam radiotherapy to the entire breast 5 days a week for 5-6 weeks.

Patients are followed at 1 month and then every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ductal carcinoma in situ or invasive adenocarcinoma of the breast

  * Primary tumor classified as T1, T2, or T3
* Candidate for breast-conserving surgery
* Must have undergone lumpectomy with negative margins or minimal margin involvement
* Currently undergoing re-excision of the biopsy cavity and/or sentinel lymph node biopsy or axillary lymph node dissection
* No evidence of metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Adult

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,500/mm^3
* Granulocyte count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* No other malignancies within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer

  * Prior contralateral breast cancer allowed if curatively treated more than 5 years previously
* No severe psychiatric or medical illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the involved breast

Surgery

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-11; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Determine the effect of intraoperative radiotherapy boost to the tumor bed on acute complications after lumpectomy (before whole breast irradiation) in women with ductal carcinoma in situ or invasive adenocarcinoma of the breast. | Patients are followed at 1 month and then every 3 months for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shelli Hanks, MD, Study Chair — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States